CLINICAL TRIAL: NCT04583267
Title: HIV Pre-exposure Prophylaxis Implementation Study in South Korea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4-2018-0671
Record Dates: First submitted 2020-09-18; First posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Emtricitabine; Racivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PrEP (Experimental)
  Interventions: Drug: tenofovir disoproxil fumarate (TDF) 300mg co-formulated with emtricitabine (FTC 200mg) once daily oral administration

INTERVENTIONS:
Drug: tenofovir disoproxil fumarate (TDF) 300mg co-formulated with emtricitabine (FTC 200mg) once daily oral administration — Participants will take tenofovir disoproxil fumarate (TDF) 300mg co-formulated with emtricitabine (FTC 200mg) once daily oral administration for preventing HIV infection.

SUMMARY:
The primary objective of this study is to examine acceptability, patterns of use, rates of adherence, safety , and measured levels of drug when high risk men who have sex with men (MSM) are provided open-label tenofovir/emtricitabine (TDF/FTC) for PrEP in South Korea. Secondary objectives are 1) to evaluate HIV incidence among study participants, 2) to evaluate risk behavior and risk compensation among study participants, and 3) to identify barriers and facilitators of PrEP among study participants. The design of this study is a prospective, open-label cohort study assessing PrEP implementation in tertiary hospital infectious diseases clinics in South Korea for 1 year. Baseline data will be collected 1 months before initiation of PrEP, and the date of initiation of PrEP. All persons receiving PrEP should be seen at 1 month since PrEP initiation and at least every 3 months to assess side effects, adherence, and HIV acquisition risk behaviors. Drug concentration will be measured every 6 months. It is anticipated that approximately 100 Korean MSM will be enrolled in this study.

DETAILED DESCRIPTION:
1. Primary Objectives

   • To examine acceptability, patterns of use, rates of adherence, safety , and measured levels of drug when high risk MSM are provided open-label TDF/FTC for PrEP in South Korea
2. Secondary Objectives

   * To evaluate HIV incidence among study participants
   * To evaluate risk behavior and risk compensation among study participants
   * To identify barriers and facilitators of PrEP among study participants
3. Study design Prospective, open-label cohort study assessing PrEP delivery in tertiary hospital infectious diseases clinics in South Korea for 1 year
4. Evaluation

   * Baseline evaluation

     1. HIV testing and the documentation of results are required to confirm that patients do not have HIV infection when they start taking PrEP medications. HIV Ag/anti HIV Ab combo assay should be performed before starting PrEP. Negative result of HIV Ag/anti HIV Ab combo assay within 1 week should be ascertained before PrEP initiation. Results from rapid test with oral specimen or unreliable testing results cannot be acknowledged.
     2. Renal function with estimated creatinine clearance (eCrCl) should be evaluated before starting TDF/FTC. TDF/FTC can be prescribed for persons with eCrCl ≥60 ml/min. Any person with an eCrCl of <60 ml/min should not be prescribed PrEP with TDF/FTC.
     3. Testing for hepatitis B virus (HBsAg, HBsAb) and hepatitis C virus (HCV Ab) should be performed before starting PrEP. Hepatitis B virus vaccination is recommended for MSM without HBsAb.
     4. Acute HIV infection must be excluded by symptom history, physical examinations and appropriate HIV testing before PrEP is prescribed.
     5. If HIV testing shows intermediate results, clinician should hold PrEP initiation, make efforts to identify symptoms and signs of acute viral infections, and do follow up HIV testing.
   * Follow up and monitoring during PrEP

     1. All persons receiving PrEP should be seen at 1 month since PrEP initiation and at least every 3 months to assess side effects, adherence, and HIV acquisition risk behaviors.
     2. All persons receiving PrEP should be seen at least every 3 months to assess for signs or symptoms of acute infection and repeat HIV testing (HIV Ag/anti HIV Ab combo assay). If acute infection is suspected, HIV RNA testing should be performed.
     3. Confirmative HIV testing (western blot assay) and HIV RNA testing should be performed for persons with positive results of screening assay (HIV Ag/anti HIV Ab assay). Resistance testing should be performed for persons with confirmed HIV infection during PrEP.
     4. If acute HIV infection is suspected during PrEP, PrEP should be stopped, combination antiretroviral therapy with TDF/FTC+boosted protease inhibitor (darunavir/ritonavir) or TDF/FTC + dolutegravir should be prescribed.
     5. All persons receiving PrEP should be seen at least every 3 months to monitor eCrCl.
     6. Sexually active persons receiving PrEP should be seen at least every 6 months to conduct tests for sexually transmitted infections (i.e. syphilis, gonorrhea, chlamydia).
     7. Assessments of bone health are not routinely recommended before the initiation of PrEP or for the monitoring of persons while taking PrEP. However, assessment for bone health can be considered for any person who has a history of pathologic fractures or who has significant risk factors for osteoporosis mineral density PrEP.
     8. All persons receiving PrEP should be seen at least 12 months to evaluate the need to continue PrEP as a component of HIV prevention considering HIV acquisition risk behavior, adherence, and so on.
5. Measurement Baseline data will be collected 1 months before initiation of PrEP, and the date of initiation of PrEP.

All persons receiving PrEP should be seen at 1 month since PrEP initiation and at least every 3 months to assess side effects, adherence, and HIV acquisition risk behaviors. During every visits including screening visit, below measures are assessed.

* Diagnostic testing: HIV testing with a fourth generation HIV Ag/Ab test, HIV RNA assay, serologic test for syphilis using VDRL or RPR, screening for gonorrhoea and chlamydia using nucleic acid amplification test
* Sociodemographics and sexual behaviors: demographic and sexual behavioral data are collected by trained interviewers using standardized questionnaires including residence, living situation, employment, insurance status, income, housing/food instability, drug use, number of anal sex partners, episodes in the past 3 months, condom use, partner HIV serostatus, sexual position, etc.

ELIGIBILITY:
Inclusion Criteria:

* MSM
* Adults
* Participants have to be HIV negative by a fourth generation HIV antigen/antibody (Ag/Ab) test
* Urine dipstick with negative or trace protein
* eGFR ≥60 mL/min
* HBsAg negative
* Condomless anal sex in the past 6 months or diagnosed with at least one STI in the past 6 months

Exclusion Criteria:

* Serious medical or psychiatric comorbidities
* Taking nephrotoxic medications
* Suspected acute HIV infection by physician

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-08-28 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Rate of adherence to PrEP with TDF/FTC | 3 months
  Rate of adherence will be measured by self report using visual analogue scale, pill counts, and drug concentration.
Rate of adherence to PrEP with TDF/FTC | 6 months
  Rate of adherence will be measured by self report using visual analogue scale, pill counts, and drug concentration.
Rate of adherence to PrEP with TDF/FTC | 9 months
  Rate of adherence will be measured by self report using visual analogue scale, pill counts, and drug concentration.
Rate of adherence to PrEP with TDF/FTC | 12 months
  Rate of adherence will be measured by self report using visual analogue scale, pill counts, and drug concentration.

SECONDARY OUTCOMES:
Number of participants with decreased eGFR | 1) 3 months, 2) 6 months, 3) 9 months, 4) 12 months
  eGFR will be calculated using the simplified modification of diet in renal disease (MDRD) equation.
Number of participants who experienced adverse events related to TDF/FTC | 1) 3 months, 2) 6 months, 3) 9 months, 4) 12 months
  data on adverse events related to TDF/FTC will be collected by questionnaire for adverse events
Rate of condom use of participants | 1) 3 months, 2) 6 months, 3) 9 months, 4) 12 months
  data on rate of condom use of participants will be collected by questionnaire for sexual behaviors of participants
Number of sexual partners of participants | 1) 3 months, 2) 6 months, 3) 9 months, 4) 12 months
  data on number of sexual partners of participants will be collected by questionnaire for sexual behaviors of participants
Incidence of sexually transmitted diseases | 1) 3 months, 2) 6 months, 3) 9 months, 4) 12 months
  laboratory tests for STD such as VDRL, FTA-ABS, and multiplex urine PCR for STD will be performed for participants. In addition, questionnaire for STD history will be performed.
Number of participants who are willing to continue PrEP | 1) 3 months, 2) 6 months, 3) 9 months, 4) 12 months
  this information will be collected by questionnaire. Visual analogue scale will be used for measuring willingness (minimum value 0, maximum value 100, higher scores mean a better willingness.)
Reasons of non-adherence to PrEP among study participants | 1) 3 months, 2) 6 months, 3) 9 months, 4) 12 months
  this information will be collected by questionnaire. Visual analogue scale will be used for measuring adherence (minimum value 0, maximum value 100, higher scores mean a better adherence)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Yong Choi, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No